CLINICAL TRIAL: NCT02547818
Title: A Phase III Safety and Efficacy Study of ALZT-OP1 in Subjects With Evidence of Early Alzheimer's Disease
Brief Title: Safety and Efficacy Study of ALZT-OP1 in Subjects With Evidence of Early Alzheimer's Disease
Acronym: COGNITE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AZTherapies, Inc. (Industry)
Collaborators: PharmaConsulting Group (Unknown); KCAS Bio (Unknown); APCER Life Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZT-001
Record Dates: First submitted 2015-09-10; First posted 2015-09-11 (Estimated); Last update posted 2021-11-10 (Actual); Status verified 2020-11

CONDITIONS: Alzheimer's Disease
Keywords: Early stage AD; MCI; aMCI; prodromal; Memory loss; Memory problems; Aging; Early Alzheimer's Disease; Early AD
MeSH Terms: conditions — Alzheimer Disease; Memory Disorders | interventions — Cromolyn Sodium; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group I (Active Comparator): ALZT-OP1a active capsules for inhalation and ALZT-OP1b placebo capsules for oral administration.
  Interventions: Drug: ALZT-OP1a; Other: Placebo ALZT-OP1b
- Group II (Active Comparator): ALZT-OP1a active capsules for inhalation and ALZT-OP1b active tablets for oral administration.
  Interventions: Drug: ALZT-OP1a; Drug: ALZT-OP1b
- Group III (Active Comparator): ALZT-OP1a placebo capsules for inhalation and ALZT-OP1b active tablets for oral administration.
  Interventions: Drug: ALZT-OP1b; Other: Placebo ALZT-OP1a
- Group IV (Placebo Comparator): ALZT-OP1a placebo capsules for inhalation and ALZT-OP1b placebo tablets for oral administration.
  Interventions: Other: Placebo ALZT-OP1a; Other: Placebo ALZT-OP1b

INTERVENTIONS:
Drug: ALZT-OP1a — 1) Mast cell stabilizer, 2) Neuroinflammatory microglial modulator, 3) A-beta oligomerization inhibitor, and 4) anti-inflammatory
  Other Names: Cromolyn
  Arms: Group I; Group II
Drug: ALZT-OP1b — Anti-inflammatory
  Other Names: Ibuprofen
  Arms: Group II; Group III
Other: Placebo ALZT-OP1a — Non-active capsules
  Arms: Group III; Group IV
Other: Placebo ALZT-OP1b — Non-active tablets
  Arms: Group I; Group IV

SUMMARY:
This is a global Phase III, randomized, double-blinded, placebo-controlled study for subjects with evidence of early AD. The protocol is designed to determine whether ALZT-OP1 combination treatment (ALZT-OP1a + ALZT-OP1b) will slow down, arrests, or reverse cognitive and functional decline, in subjects with evidence of early stage Alzheimer's disease (AD).

DETAILED DESCRIPTION:
This Phase III study is designed as a randomized, double-blinded, placebo-controlled study for subjects with evidence of early AD. The study will evaluate safety and tolerability, efficacy as measured by CDR-SB, and will determine if the combination therapy ALZT-OP1 will slow down, arrests, or reverse cognitive and functional decline in an early stage AD population.

Subjects will be randomly assigned to one of four treatment arms: Group I will consist of ALZT-OP1a (cromolyn) for inhalation, plus an oral placebo tablet; OR the Group II arm, which will consist of ALZT-OP1 combination therapy ALZT-OP1a (cromolyn) for inhalation, plus ALZT-OP1b (ibuprofen) tablet for oral administration; OR to the Group III arm, which will consist of inhaled placebo, plus ALZT-OP1b (ibuprofen) tablet for oral administration; OR to the Group IV placebo arm, which will consist of inhaled placebo plus an oral placebo tablet.

A minimum of 400 evaluable subjects will be randomized to receive one of four possible treatment assignments containing various combinations of active study drug or placebo.

To account for subject dropouts (estimated rate of 30%), it is anticipated that up to 600 (or 150 subjects per treatment arm) may be recruited and randomized, to achieve a minimum of 100 evaluable subjects per treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* 55-79 years old;
* ≥ 8 years of education;
* Study partner is available who has frequent contact with the participant (e.g. an average of 10 hours per week or more), and can accompany the participant to all clinic visits for the duration of the protocol;
* Evidence of early AD, as defined by all of the following:

  1. Memory complaint by subject or study partner that is verified by a study partner;
  2. Objective memory impairment for age, documented by scoring below the education adjusted cutoff of the Logical Memory II subscale (Delayed Paragraph Recall) from the Wechsler Memory Scale Third Edition (the maximum score is 25):

     * ≤ 8 for 16 or more years of education, or
     * ≤ 4 for 8-15 years of education;
     * Essentially preserved general cognitive function;
     * Largely intact functional activities;
     * Not demented;
* Cerebrospinal fluid (CSF) biomarker results consistent with early AD, including CSF Aβ-42 levels ≥ 180 pg/mL and ≤ 690 pg/mL;
* Clinical Dementia Rating (Global) = 0.5; Memory Box score must be at least 0.5;
* Must be fluent in the language of the cognitive testing material being administered;
* Stability of permitted medications for 4 weeks prior to study start; subjects receiving acetylcholinesterase inhibitors and/or memantine should be on stable dose of those medications for at least 12 weeks prior to study start with every effort to maintain stable dose for the duration of the study;
* Visual and auditory acuity adequate for neuropsychological testing;
* Good general health with no diseases expected to interfere with the study;
* Must provide written informed consent for APOe4 genotype testing;
* Must provide written informed consent for CSF sampling.

Exclusion Criteria:

* Any significant neurological disease other than suspected incipient AD, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities;
* Major depressive episode, as described in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) within the past 6 months, which could lead to difficulty complying with the protocol;
* History of schizophrenia or bipolar disorder (DSM-IV criteria);
* History of alcohol or substance abuse or dependence within the past 3 years (DSM-IV criteria);
* Currently taking medications that could lead to difficulty complying with the protocol; subjects must be on a stable dose of current medications for 4 weeks prior to study entry, with the exception of acetylcholinesterase inhibitors and/or memantine, which must be on a stable dose for at least 12 weeks prior to study entry;
* Investigational agents are prohibited one month prior to entry and for the duration of the trial;
* Currently taking medications known to be CYP2C9 inducers (i.e. carbamazepine and rifampicin);
* Currently taking cromolyn, or have taken cromolyn, within the past 12 months;
* Chronic daily use of high-dose NSAID for osteoarthritis, rheumatoid arthritis, or other chronic inflammatory diseases ("chronic" defined as 3200 mg/day for >2 weeks);
* Chronic daily use of aspirin exceeding standard of care guidelines for low dose aspirin therapy for prevention of stroke and/or other recommended uses;
* Allergy to cromolyn (also known as Intal®, Nasalcrom®, Opticrom®, Gastrocrom®, etc.);
* Allergies to ibuprofen (Advil®, Motrin®, Nuprin®, etc.) or aspirin;
* Clinically significant respiratory disorders with impaired respiratory effort or difficulty taking inhaled drugs;
* Uncontrolled chronic asthma;
* Abnormal pulmonary function test, defined for this protocol as: FEV1/FVC < predicted value for subject AND FEV1 < 70% of predicted value, indicating moderate or severe respiratory obstruction;
* Taking inhaled protein products on a chronic basis;
* Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol;
* Pregnancy or lactation for female subjects of child-bearing potential (i.e., < two years post-menopausal or not surgically sterile);
* For sexually active male subjects, unwillingness or incapability of using appropriate contraception methods;
* Severe renal or hepatic impairment.

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Clinical Dementia Rating-Sum of Boxes (CDR-SB) | Baseline and Week 72
  The combination active treatment group will be compared to each of the single component groups, including the placebo group, the mean change from Baseline to Week 72 will be quantified.

SECONDARY OUTCOMES:
Number of Treatment Emergent Adverse Events (TEAE) | 72 weeks
  Safety will be evaluated based on the number, type, and frequency of treatment emergent adverse events. They will be individually presented for all subjects in data listings, and summarized in tables by treatment group and by treatment assignment. The AE's will be summarized and reported collectively based on information obtained through physical examination, ECG, and laboratory findings captured after dosing is initiated.

CONTACTS AND LOCATIONS:
Overall Officials: David R. Elmaleh, PhD, Study Director — AZTherapies, Inc.
Locations (121):
- United States (69):
  - Cognitive Clinical Trials, Gilbert, Arizona
  - Xenoscience, Phoenix, Arizona
  - Cognitive Clinical Trials, Scottsdale, Arizona
  - Territory Neurology & Research Institute, Tucson, Arizona
  - Alliance Research Center, Laguna Hills, California
  - Renew Behavioral Health, Long Beach, California
  - Excell Research, Inc., Oceanside, California
  - University of California Irvine School of Medicine, Orange, California
  - Asclepes Research Center, Panorama City, California
  - Artemis Clinical Research, Riverside, California
  - CITrials, Riverside, California
  - Northern California Research, Sacramento, California
  - Syrentys Clinical Research, Santa Ana, California
  - Mile High Research Center, Denver, Colorado
  - TOPAZ Clinical Research, Apopka, Florida
  - Parkinson's Disease & Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Bradenton Research Center, Bradenton, Florida
  - Finlay Medical Research Group, Greenacres City, Florida
  - Galiz Clinical Research, Hialeah, Florida
  - The Neurology Research Group, Miami, Florida
  - Premier Clinical Research Institute, Miami, Florida
  - Finlay Medical Research Group, Miami, Florida
  - Next Phase Research Alliance - Cano Health, Miami, Florida
  - IMIC, Inc., Miami, Florida
  - Next Phase Research Alliance - MetroMed, Miami, Florida
  - Next Phase Research Alliance, Miami, Florida
  - Panax, Miami Lakes, Florida
  - CNS Healthcare, Orlando, Florida
  - Pines Care Research Center, Pembroke Pines, Florida
  - Neurostudies, Inc., Port Charlotte, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Axiom Clinical Research, Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Columbus Research & Wellness Institute, Columbus, Georgia
  - Behavioral Health Care Associates, Schaumburg, Illinois
  - Eastern Maine Medical Center, Bangor, Maine
  - Coastal Health Care, Freeport, Maine
  - Samuel and Alexia Bratton Memory Clinic, Easton, Maryland
  - ActivMed Practices & Research, Inc., Methuen, Massachusetts
  - The Alzheimer's Disease Center, Quincy, Massachusetts
  - Bronson Neurobehavioral Health, Paw Paw, Michigan
  - Cognitive Clinical Trials, Bellevue, Nebraska
  - Cognitive Clinical Trials, Omaha, Nebraska
  - ActivMed Practices & Research Inc., Portsmouth, New Hampshire
  - Memory Enhancement Center of America, Eatontown, New Jersey
  - AdvancedMed Research, Lawrenceville, New Jersey
  - The NeuroCognitive Institute, Mount Arlington, New Jersey
  - Albuquerque Neuroscience, Albuquerque, New Mexico
  - Adirondack Medical Research Center, Glens Falls, New York
  - Manhattan Behavioral Medicine, New York, New York
  - Medical Research Network, New York, New York
  - Nathan S. Kline Institute for Psychiatric Research, New York, New York
  - Winifred Masterson Burke Medical Research Institute, White Plains, New York
  - ANI Neurology, PLLC Alzheimer's Memory Center, Charlotte, North Carolina
  - Raleigh Neurological Associates, Raleigh, North Carolina
  - PMG Winston-Salem, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Insight Clincial Trials, Shaker Heights, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Tulsa Clinical Research, Inc., Tulsa, Oklahoma
  - Pearl Clinical Research, Norristown, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Palmetto Health, Columbia, South Carolina
  - Metrolina Neurological Associates, PA, Rock Hill, South Carolina
  - CNS Healthcare, Memphis, Tennessee
  - Neurology Associates of Arlington, P.A., Mansfield, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Kingfisher Cooperative, Spokane, Washington
- Australia (7):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - KaRa Institute of Neurological Diseases, Macquarie Park, New South Wales
  - Pacific Private Clinic, Southport, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Geelong Private Medical Centre, Geelong, Victoria
  - Austin Health, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Bulgaria (5):
  - UMBAL "Dr. Georgi Stranski" EAD, Pleven
  - MHAT "Central Onco Hospital" Ltd., Plovdiv
  - MBAL Ruse AD, Rousse
  - "First MHAT - Sofia" EAD, Sofia
  - University Multiprofile Hospital for Active Treatment "Aleksandrovska" EAD, Sofia
- Canada (10):
  - Medical Arts Health Research, Penticton, British Columbia
  - Medical Arts Health Research, West Vancouver, British Columbia
  - Okanagan Clinical Trials, Kelowna, Britsh Columbia
  - Montreal Neurological Research Institute, Québec, Montreal
  - True North Clinical Research, Halifax, Nova Scotia
  - True North Clinical Research, Kentville, Nova Scotia
  - JBN Medical, Burlington, Ontario
  - Chatham-Kent Clinical Trials, Chatham, Ontario
  - The Centre for Memory and Aging, East York, Ontario
  - Cliniuqe de la Memoire de l'Outouais, Gatineau, Quebec
- Czechia (13):
  - Neurosanatio, s.r.o., Litomyšl, Czech Republic
  - Neurologie MU - Ondrej Koci, s.r.o., Nový Bor, Czech Republic
  - CT Center MaVfe, s.r.o, Olomouc, Czech Republic
  - Vestra Clinics, s.r.o., Rychnov nad Kněžnou, Czech Republic
  - NEUROHK, s.r.o., Choceň
  - Clinline Services s.r.o., Hostivice
  - Psychiatricka ambulance, Hradec Králové
  - Psychiatricka ambulance Supervize s.r.o., Kutná Hora
  - Krajska nemocnice Liberec a.s., Liberec
  - A-shine, s.r.o., Pilsen
  - Clintrial.s.r.o., Prague
  - Fakultni nemocnice v Motole Neurologicka klinika 2.LF UK a FN Motol, Prague
  - INEP medical s.r.o., Prague
- Hungary (5):
  - Neurologia Klinika Semmelweis Egyetem, Budapest
  - Orszagos Klinikai Idegtudomanyi Intezat, Budapest
  - Vaszary Kolos Korhaz, Esztergom
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Bekes Megyei Pandy Kalman Korhaz, Gyula
- Poland (12):
  - Cermed Pawel Hernik, Bialystok
  - Podlaskie Centrum Psychogeriatrii, Bialystok
  - Przychondnia Srodmiescie, Bydgoszcz
  - Centrum Medyczne KERMED, Bydgoszcz
  - Szpital Powiatowy w Czeladzi, Czeladź
  - Centrum Zdrowia Psychicznego Biomed - Jan Latala, Kielce
  - Centrum Medyczne Plejady, Krakow
  - Centrum Opieki Zdrowotnej Orkan-Med, Ksawerów
  - Centrum Medyczne im. Dr Karola Jonschera w Lodzi, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie, Lublin
  - CRC Sp. Zo.o., Poznan
  - Euromedis Sp. Zo.o, Szczecin